CLINICAL TRIAL: NCT06929507
Title: The Impact of Intravitreal Injection of Anti-vascular Endothelial Growth Factor Faricimab on Renal Function in Patients With Diabetes Mellitus
Brief Title: Impact of Intravitreal Faricimab on Renal Function in Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Alexandroupolis (Other)
Responsible Party: Principal Investigator, Asli Perente, Consultant Ophthalmologist, University Hospital, Alexandroupolis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12808/10-03-2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-16 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Renal Function Disorder; Diabetic Macular Edema (DME); Neovascular Age Related Macular Degeneration
Keywords: renal function; intravitreal injection of anti-VEGF; faricimab; diabetic macular edema; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who will be treated with intravitreal injections of Faricimab (Active Comparator): Diabetic patients with either diabetic macular edema (DME) or neovascular age related macular degeneration (nAMD) who will be treated with intravitreal injection of Faricimab.
  Interventions: Drug: Intravitreal injection of Faricimab or Aflibercept 2 mg
- Patients who will be treated with intravitreal injections of Aflibercept 2 mg (Active Comparator): Diabetic patients with either diabetic macular edema (DME) or neovascular age related macular degeneration (nAMD), or macular edema secondary to retinal vein occlusion who will be treated with intravitreal injection of Aflibercept 2 mg.
  Interventions: Drug: Intravitreal injection of Faricimab or Aflibercept 2 mg

INTERVENTIONS:
Drug: Intravitreal injection of Faricimab or Aflibercept 2 mg — Anti-VEGF agents Faricimab (Vabysmo) or Aflibercept 2 mg (Eylea) will be delivered intravitreally
  Other Names: Vabysmo; Eylea

SUMMARY:
This study aims to investigate the impact of intravitreal injection of anti-vascular endothelial growth factor (anti VEGF) Faricimab on renal function of diabetic patients. Faricimab is a new anti-VEGF drug which inhibits both VEGF-A and Ang-2 and it is used for the treatment of diabetic macular edema and neovascular age related macular degeneration. It is known that previous anti-VEGF agents has systematic absorption and may cause deterioration in renal function of the patients. However, the effect of Faricimab on kidney function has not been investigated yet. Taking into account that Ang-2 has destructive effect on kidneys, the investigation of the effect of its inhibition in diabetic patients who have already renal function deterioration may provide a valuable information in scientific community.

DETAILED DESCRIPTION:
For the purposes of this study, 60 diabetic patients who need intravitreal injections of anti-VEGF for either diabetic macular edema or neovascular age related macular degeneration will be enrolled. 30 patients will consist the study group and they will receive Faricimab and the remaining 30 patients will receive Aflibercept 2 mg. Before the initiation of therapy, laboratory tests including HbA1c, eGFR, plasma creatinine, urine albumin to urine creatinine ratio (ACR) will be ordered to investigate the glycemic control and the renal function of the patients.The best corrected visual acuity (BCVA), the intraocular pressure (IOP) and the anterior segments will be assessed on each visit. The optical coherence tomography (OCT) will be used for the assessment of centra macular thickness (CMT). The results will be assessed at baseline and then at 6 months and 12 months from the initiation of therapy. The statistical analysis will be performed at the end of study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes
* Patients with DME or nAMD or macular edema secondary to retinal vein occlusion
* Patients already receiving nephroprotective drugs

Exclusion Criteria:

* Patients with end stage renal disease
* Pregnancy
* Patients with other retinal disorders
* Previous renal transplantation Patients under hemodialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
eGFR | 12 months
  The eGFR before the initiation of treatment and at 6 and 12 months after
ACR ration | 12 months
  The ACR ratio before the initiation of treatment and 6 and 12 months after

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - University Hospital of Alexandroupolis, Alexandroupoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shye M, Hanna RM, Patel SS, Tram-Tran N, Hou J, Mccannel C, Khalid M, Hanna M, Abdelnour L, Kurtz I. Worsening proteinuria and renal function after intravitreal vascular endothelial growth factor blockade for diabetic proliferative retinopathy. Clin Kidney J. 2020 Jun 28;13(6):969-980. doi: 10.1093/ckj/sfaa049. eCollection 2020 Dec. PMID 33391740
- [Background] Fang YC, Lai IP, Lai TT, Chen TC, Yang CH, Ho TC, Yang CM, Hsieh YT. Long-Term Change in Renal Function After Intravitreal Anti-VEGF Treatment for Diabetic Macular Edema: A 2-Year Retrospective Cohort Study. Ophthalmol Ther. 2023 Dec;12(6):2977-2988. doi: 10.1007/s40123-023-00771-4. Epub 2023 Aug 17. PMID 37589931
- [Background] Li M, Popovic Z, Chu C, Reichetzeder C, Pommer W, Kramer BK, Hocher B. Impact of Angiopoietin-2 on Kidney Diseases. Kidney Dis (Basel). 2023 Mar 14;9(3):143-156. doi: 10.1159/000529774. eCollection 2023 May. PMID 38306230